CLINICAL TRIAL: NCT06325085
Title: Combined Effects of Restorative and Compensatory Rehabilitation Techniques on Executive Functions in Stroke With Mild Cognitive Impairment
Brief Title: Compensatory and Restorative Rehabilitation Techniques in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ayesha Saddiqa
Record Dates: First submitted 2024-03-17; First posted 2024-03-22 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Cognitive Impairment
Keywords: Compensatory rehabilitation; Restorative Rehabilitation; Cognition; Stroke; Executive Functioning
MeSH Terms: conditions — Cognitive Dysfunction; Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Compensatory and restorative rehabilitation techniques (Experimental): compensatory and restorative rehabilitation techniques in stroke patients
  Interventions: Other: compensatory and restorative rehabilitation techniques
- Traditional cognitive Rehabilitation training (Active Comparator): Naming words Counting numbers backwards Spell the word backwards
  Interventions: Other: Traditional cognitive rehabilitation training

INTERVENTIONS:
Other: compensatory and restorative rehabilitation techniques — compensatory and restorative rehabilitation techniques Frequency: 10 reps 2-3 times/week for 3 consecutive weeks then evaluation of the effects.
  Continue the same techniques for 3 more weeks and then evaluate the retention effects of restorative and compensatory rehabilitation techniques will be evaluated by 9th week.
  Arms: Compensatory and restorative rehabilitation techniques
Other: Traditional cognitive rehabilitation training — Naming words ( ask patient to name food, states, family members) Counting numbers backwards, backward counting of days and months) Spell the word backwards, remembering a piece of information Frequency: 10 reps 2-3 times/week for 3 consecutive weeks then evaluation of the effects.
  Continue the same techniques for 3 more weeks and then evaluate the retention effects of restorative and compensatory rehabilitation techniques will be evaluated by 9th week.
  Arms: Traditional cognitive Rehabilitation training

SUMMARY:
The aim of this randomized controlled trial is to find the combined effects of restorative and compensatory cognitive rehabilitation techniques in mild cognitive impairment after stroke.

DETAILED DESCRIPTION:
Stroke is a prevalent medical neurological condition that often results in cognitive impairments, particularly in the domain of executive functions. Cognitive impairment has a significant impact on executive function in stroke subjects. Cognitive impairment on the stroke survivor exist on any single domain such as attention, spatial ability, language and executive ability more frequently than the multiple domains.

Cognitive training has been shown to be beneficial for rehabilitation of patients with cognitive impairment, but the underlying mechanisms remain unclear.

The combination of restorative and compensatory rehabilitation techniques is beneficial for gaining control over cognitive rehabilitation techniques will improve executive functions. The retention effects evaluated additionally will add a broad insight in this regard. It will improve the learning power of brain through neural plasticity. This leads to restoration of everyday functioning. This study aims to investigate the effects of two distinct rehabilitation approaches on the executive functions of stroke survivors with MCI. Understanding how these rehabilitation strategies impact cognitive recovery is essential for individuals living with post-stroke cognitive impairments.

ELIGIBILITY:
Inclusion Criteria:

* Age between 50 and 70 years
* Both Genders
* Individuals diagnosed with stroke 6 months before enrollment
* Minimum 6 years of schooling
* Patients with mild cognitive impairment (score 18-25 on MOCA)
* Individuals able to maintain sitting and standing balance (score 41 on berg balance scale)

Exclusion Criteria:

* >10 on post stroke depression rating scale (PSDRS)
* Spasticity (>3 on Ashworth scale)
* Other psychological disorders
* Patients diagnosed with Alzheimer's and dementia

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-04-16 (Actual); Primary Completion 2025-08-28 (Actual); Study Completion 2025-08-29 (Actual)

PRIMARY OUTCOMES:
Montreal cognitive assessment test (Urdu version) | 6 weeks
  MOCA assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuo-constructional skills, conceptual thinking and orientation. The test is one page,30 point test that can be administered in 10 minutes. MOCA is scored by obtaining an item total and the author recommend a clinical cutoff score of 26.is a Patient-completed, condition-specific functional status questionnaire with 10 items including pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping and recreation.
Cognitive assessment scale for stroke patients (CASP) | 6 weeks
  Its a rapid test for screening post stroke cognitive impairment. It can be performed at the patient bedside by a non expert examiner. A CASP score of 35/36 should alert to possible presence of cognitive impairment. Score can help predict medium level cognitive impairment.

SECONDARY OUTCOMES:
Stroke specific quality of life questionnaire (Urdu version) | 6 weeks
  The SS-QOL questionnaire assesses health related quality of life specific to stroke survivors covering almost 12 domains
Modified Rankin Scale (MRS) | 6 weeks
  It measures degree of disability or dependence in daily activities of people who have suffered stroke or other neurological disability. It is one of the most widely used clinical patients are graded

CONTACTS AND LOCATIONS:
Overall Officials: Aroosa Tariq, MS-NMPT, Principal Investigator — Riphah International University
Locations (1):
- Shafi Hospital Dina, Dina, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No